CLINICAL TRIAL: NCT03805165
Title: Associations of Nighttime Light Exposure During Pregnancy With Neonatal Jaundice：a Multi-centre Prospective Study in China
Acronym: jaundice
Status: Completed | Type: Observational
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yang jie, Director of neonatology of GuangdongWCH, Guangdong Women and Children Hospital
Other Study IDs: Guangdong WCH
Record Dates: First submitted 2018-12-25; First posted 2019-01-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Jaundice, Neonatal
Keywords: nighttime light exposure ，neonatal jaundice，China
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neonate: transcutaneous bilirubin(TCB) measurements were performed with 2977 neonates at designated time points. The mean NTL exposure during pregnancy was respectively calculated based on each participant's residential address over the study course.

SUMMARY:
Make a neonatal jaundiced nomogram on Chinese jaundice data by joinning the major neonate centers all around China.

DETAILED DESCRIPTION:
This was a multi-centre prospective study. All infants included were born in 8 hospitals in the southern, eastern, northern, western and central regions of mainland China in 2019. A total of 20839 transcutaneous bilirubin(TCB) measurements were performed with 2977 neonates at designated time points. The mean NTL exposure during pregnancy was respectively calculated based on each participant's residential address over the study course. The primary outcome was whether the neonate was diagnosed with hyperbilirubinemia within the first seven days of life. The effect of maternal nocturnal light exposure on neonate jaundice analyzed with lasso regression and random forest machine learning methods.

ELIGIBILITY:
Inclusion Criteria:

gestational age more than 35 weeks(≥35) -

Exclusion Criteria:

all kinds of congenital diseases, infants with pathologic jaundice

-

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and near term newborns, whos gestational age was more than 35 weeks(≥35)
Sampling Method: Probability Sample
Enrollment: 2977 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Hour-specific Transcutaneous Bilirubin Level | 1 year
  make neonatal jaundiced nomogram base on the hour-specific transcutaneous bilirubin data
whether the neonate was diagnosed with hyperbilirubinemia within the first seven days of life | 2019
  whether the neonate was diagnosed with hyperbilirubinemia within the first seven days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China